CLINICAL TRIAL: NCT00008788
Title: Osteoporosis in Children and Adults Following Liver Transplantation
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Center for Research Resources (NCRR) (NIH)
Other Study IDs: NCRR-M01RR00400-0664
Record Dates: First submitted 2001-01-16; First posted 2001-01-18 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-12

CONDITIONS: Osteoporosis; Liver Transplantation
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Cross-Sectional

SUMMARY:
This pilot project aims to 1) estimate the prevalence of osteoporosis in adults having undergone liver transplantation in childhood, and 2) identify risk factors for osteoporosis in this group. We aim to study 40 individuals.

DETAILED DESCRIPTION:
Background: Osteoporosis is defined as an absolute decrease in the amount of bone (volume and/or density). Chronic liver disease is associated with osteoporosis in both adults and children. Bone density is also decreased in the months immediately after liver transplantation, but improves to pretransplant values after 1 to 2 years. Immunosuppressive agents, most notably steroids, are a cause of osteoporosis. However, studies on adults have shown that bone densities afer transplantation continue to improve within the normal range for healthy adults. In the case of children, bone accretion is necessary for growth. Chronic liver disease and transplantation in childhood will have an adverse effect on bone metabolism and the outcome in terms of bone density after the growth period cannot be predicted on individuals transplanted as adults or other transplant groups.

ELIGIBILITY:
* Liver transplantation in childhood or young adulthood

Ages: 16 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States